CLINICAL TRIAL: NCT02749786
Title: Expansion Arm of Papulopustular Rosacea Gene Expression Profiling to Include Normal Individuals as Anatomic Site Specific Controls
Brief Title: Genetic Basis of Rosacea Study (Control)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Anne Chang, Associate Professor of Dermatology, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 22419
Record Dates: First submitted 2016-04-18; First posted 2016-04-25 (Estimated); Last update posted 2019-09-26 (Actual); Status verified 2019-09

CONDITIONS: Rosacea
MeSH Terms: conditions — Rosacea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Control Group (Other): Participants who do not have rosacea (control group)
  Interventions: Other: Skin Biopsy

INTERVENTIONS:
Other: Skin Biopsy — Skin biopsies will be performed via the Keys punch technique from normal facial skin.

SUMMARY:
Rosacea is a common disease characterized by inflammation and vascular abnormalities of the facial skin and ocular surface. It it considered to be a syndrome encompassing various combinations of cutaneous signs including flushing, erythema, telangiectasia, papules, edema, ocular lesions, and rhinophyma. The exact etiology of cutaneous rosacea is unknown but is characterized by persistent vasodilation, increased vascular permeability, and vascular hyper-reactivity of the microcirculation of the central part of the face. The purpose of this study is to develop gene expression profiles of papulopustular rosacea compared to those of normal skin. The investigator hopes to better understand the abnormal gene functions that might contribute to this condition. This understanding may lead to the development of additional and better treatments for rosacea.

ELIGIBILITY:
Inclusion criteria include:

1. Fitzpatrick skin type II or III
2. Age greater than or equal to 18 years
3. Individuals without a history of rosacea

Exclusion criteria include:

1. Women who are pregnant or lactating
2. Use of topical prescription medications or procedures to the face within one month of enrollment
3. Skin conditions that might interfere with interpretation of procedure results (at the discretion of the investigator)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-01-21 (Actual); Primary Completion 2016-08-01 (Actual); Study Completion 2016-08-01 (Actual)

PRIMARY OUTCOMES:
Gene expression profile of papulopustular rosacea compared to normal skin and skin from individuals without rosacea. | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Anne Chang, Principal Investigator — Stanford University
Locations (1):
- Stanford Dermatology, Redwood City, California, United States

IPD SHARING:
Plan to Share IPD: No